CLINICAL TRIAL: NCT00303251
Title: A Phase I/II Dose Escalating Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of TKI258 (CHIR-258) in Patients With Locally Advanced or Metastatic Melanoma
Brief Title: Safety of TKI258 in Advanced/Metastatic Melanoma Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2105
Record Dates: First submitted 2006-03-14; First posted 2006-03-16 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2013-02

CONDITIONS: Melanoma
Keywords: Locally Advanced or Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

ARMS (1):
- TKI258 (Experimental)
  Interventions: Drug: TKI258

INTERVENTIONS:
Drug: TKI258

SUMMARY:
This study is an open-label, dose-escalating study to delineate the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of TKI258. Pharmacokinetics and pharmacodynamics will be performed on all subjects. The eligible subject population consists of subjects who have been diagnosed with locally advanced or metastatic melanoma that is refractory to standard therapy or for which no curative standard therapy exists.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of locally advanced or metastatic melanoma (American Joint Committee on Cancer [AJCC] stage IIIB, IIIC or IV) that is refractory to standard therapy or for which no curative standard therapy exists.
* Measurable disease
* Must be eighteen years of age or older
* Must meet baseline laboratory requirements
* ECOG performance status 0 or 1
* Adults of reproductive potential must agree to use effective contraception or be sterile

Exclusion Criteria:

* Concurrent therapy with any other investigational agent
* Uncontrolled central nervous system metastases
* Impaired cardiac function or clinically significant cardiac disease
* Received

  * chemotherapy, targeted therapy or monoclonal antibody therapy ≤4 weeks
  * biological therapy or immunotherapy (therapeutic or diagnostic) ≤2 weeks
  * an investigational agent (therapeutic or diagnostic) ≤4 weeks prior to starting study drug or has not recovered from side effects of such therapy
* Received any hematopoietic colony-stimulating factor (e.g., G-CSF, GM-CSF) ≤ 2 weeks prior to starting study drug. Erythropoietin is allowed.
* Has undergone major surgery ≤ 2 weeks prior to starting study drug or has not recovered from side effects of such surgery.
* Malabsorption syndrome or uncontrolled gastrointestinal symptoms such as nausea, diarrhea, vomiting
* Pregnant or breast feeding women
* History of another primary malignancy that is currently clinically significant or currently requires active intervention.
* Chronic anticoagulation therapy with full strength aspirin, Coumadin, or heparin.
* History of thromboembolic or cerebrovascular events within the last 12 months.
* History of rectal bleeding, bloody vomit, or spitting up blood within the last 3 months.
* Known diagnosis of HIV infection (HIV testing is not mandatory)
* Use of ketoconazole, erythromycin, carbamazepine, phenobarbital, phenytoin, rifampin, St. John's wort and quinidine is prohibited.
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study-drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, make the patient inappropriate for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-04; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Dose Expansion: Determine the maximum tolerated dose based on dose limiting toxicity of TKI258 | end of dose escalation
Dose Expansion: Determine the plasma and whole blood pharmacokinetics of orally administered TKI258 | PK run-in days 1 & 2, cycle 1 days 1, 8, 15, 16, 28, cycle 2 day 15, cycle 2+ day 28
Dose Escalation: Assess tumor response according to RECIST as measured by response rate and lack of early progressive disease (<=2 months) | every 8 weeks

SECONDARY OUTCOMES:
Assess the safety profile of TKI258 in this patient population | PK run in day 1 & 2, cycle 1 day 8, 15, 28, cycle 2+ day 15 & 28, end of study
Assess the effect of TKI258 on biomarkers in the blood | PK run day 1 & 2, cycle 1 day 2, 15, 28, cycle 2+ day 28, end of study
Assess biomarker changes in tumor/nevi biopsies and archival tumor tissues where accessible, pre- and post-treatment | baseline, cycle 1 day 15, end of study
Assess changes in tumor glucose metabolism/cell viability between pre- and post-treatment using [18F]-FDG-PET | baseline, cycle 1 day 15, cycle 2 day 28
Assess anti-angiogenic effects of TKI258 using DCE-MRI pre- and post-treatment | baseline, cycle 1 day 2 and cycle 2 day 28

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - MD Anderson Cancer, Houston, Texas

REFERENCES:
- [Derived] Wang X, Kay A, Anak O, Angevin E, Escudier B, Zhou W, Feng Y, Dugan M, Schran H. Population pharmacokinetic/pharmacodynamic modeling to assist dosing schedule selection for dovitinib. J Clin Pharmacol. 2013 Jan;53(1):14-20. doi: 10.1177/0091270011433330. Epub 2013 Jan 24. PMID 23400739
- [Derived] Kim KB, Chesney J, Robinson D, Gardner H, Shi MM, Kirkwood JM. Phase I/II and pharmacodynamic study of dovitinib (TKI258), an inhibitor of fibroblast growth factor receptors and VEGF receptors, in patients with advanced melanoma. Clin Cancer Res. 2011 Dec 1;17(23):7451-61. doi: 10.1158/1078-0432.CCR-11-1747. Epub 2011 Oct 5. PMID 21976540
- See also: Results for (Study ID) from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4202